CLINICAL TRIAL: NCT01349374
Title: Study Aiming to Collect Skin Samples of Diabetic Patients and Healthy Volunteers for Cellular Reprogramming, Within the Framework of New Therapeutic Strategies in Diabetes Treatment
Brief Title: Skin Samples of Diabetic Patients and Healthy Volunteers Collection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2010-A01127-32
Record Dates: First submitted 2011-05-03; First posted 2011-05-06 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2011-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group1 (Experimental): healthy volunteers
  Interventions: Other: skin biopsy
- group2 (Experimental): Unaffected siblings of MODY patients
  Interventions: Other: skin biopsy
- Group3 (Experimental): Type2 Diabetic patients
  Interventions: Other: skin biopsy
- Group4 (Experimental): MODY patients
  Interventions: Other: skin biopsy

INTERVENTIONS:
Other: skin biopsy — Obtention of skin micro-samples collected from healthy volunteers and diabetic patients (type 2 and MODY), intended to be used afterwards to obtain stem cell lines, in the framework of new therapeutic strategies of type 2 diabetes.

SUMMARY:
The main objective of this study is the Obtention of skin micro-samples collected from healthy volunteers and diabetic patients (type 2 and MODY), intended to be used afterwards to obtain stem cell lines, in the framework of new therapeutic strategies of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients diagnosed for type 2 diabetes, with a BMI between 20 and 25, without familial history and known genetic cause of diabetes.
* Diabetic patients diagnosed for MODY diabetes (1, 2, 3, 4, 5 or 6), with a BMI between 20 and 25.
* Healthy volunteers, siblings of MODY patients (1, 2, 3, 4, 5 or 6).
* Healthy volunteers without familial history of diabetes.
* Patients over 18 years old.
* Patients with social insurance coverage
* Patients who signed a consent form

Exclusion Criteria:

* Type 1 diabetic patients.
* Pregnant women or women who might get pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Nothing will be measured, the aim of the study is the obtention of skin micro-samples collected from healthy volunteers and diabetic patients (type 2 and MODY), intended to be used afterwards to obtain stem cell lines. | patients will be followed for the duration of hospital stay, an expected average of 2 hours.
  * Each patient will have a consultation at the hospital. During this consultation, if the patient agrees to participate in the study, the doctor will make him/her sign a consent form and an appointment will be scheduled with the dermatologist for the skin biopsy.
  * The dermatologist will perform the skin biopsy, the sample will then be carried to the Evry genopole, where the derivation of dermal fibroblasts will be done, and the cells will then be sent to iPierian center, in California, which will take care of the obtention of cell lines.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France